CLINICAL TRIAL: NCT04029038
Title: Phase I/II Study of Dual CD19-CD22 Chimeric Antigen Receptor (CAR) T Cells in Patients With Advanced CD19+ CD22+ Lymphoid Malignancies
Brief Title: Modified Immune Cells (CD19-CD22 CAR T Cells) in Treating Patients With Recurrent or Refractory CD19 Positive, CD22 Positive Leukemia or Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0042; NCI-2019-04229 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0042 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: CD19 Positive; CD22 Positive; Minimal Residual Disease; Progressive Disease; Recurrent B Acute Lymphoblastic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Non-Hodgkin Lymphoma; Refractory B Acute Lymphoblastic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Neoplasm, Residual; Disease Progression; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CD19-CD22 CAR T cells) (Experimental): Patients receive standard of care cyclophosphamide IV over 30 minutes and fludarabine IV over 30 minutes on days -5, -4, and -3, and then receive CD19-CD22 CAR T cells IV on day 0. Patients with relapsed or persistent disease after a protocol assessment may receive a second infusion of CD19-CD22 CAR T cells.
  Interventions: Biological: Autologous CD19/CD22 Chimeric Antigen Receptor T-cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Autologous CD19/CD22 Chimeric Antigen Receptor T-cells — Given IV
  Other Names: Autologous Anti-CD19/CD22 CAR-T Cells; Autologous CD19/CD22 CAR T Cells; Autologous CD19/CD22 CAR T-cells; Autologous CD19/CD22 Chimeric Antigen Receptor T Cells
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa

SUMMARY:
This phase I/II trial studies the side effects and best dose of modified immune cells called CD19-CD22 chimeric antigen receptor (CAR) T cells in treating patients with CD19 positive(+), CD22+ B-acute lymphoblastic leukemia, chronic lymphocytic leukemia, or non-Hodgkin's lymphoma that has come back (recurrent) or does not respond to treatment (refractory). T-cells are collected from the patient and genetic materials called "chimeric antigen receptors (CAR)" are transferred to the collected T-cells. The CAR T-cells are then infused back to the patient's body. Giving CD19- CD22 CAR T cells after chemotherapy may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of infusion with chimeric antigen receptor T cells targeting CD19 and CD22.

II. To find the recommended phase II dose for recurrent/refractory CD19+CD22+ B cell malignancies.

SECONDARY OBJECTIVES:

I. To describe the overall response rate and complete response rate of relapsed B cell malignancies treated with CAR-T cells targeting CD19 and CD22.

II. To assess other response variables including minimal residual disease (MRD) negative remission, overall survival (OS), and event free survival (EFS).

EXPLORATORY OBJECTIVES:

I. To evaluate the immune reconstitution and persistence of CAR T cells for one year post infusion.

OUTLINE: This is a phase I, dose escalation study of autologous CD19/CD22 chimeric antigen receptor T-cells (CD19-CD22 CAR T cells) followed by a phase II study.

Patients receive standard of care cyclophosphamide intravenously (IV) over 30 minutes and fludarabine IV over 30 minutes on days -5, -4, and -3, and then receive CD19-CD22 CAR T cells IV on day 0. Patients with relapsed or persistent disease after a protocol assessment may receive a second infusion of CD19-CD22 CAR T cells.

After completion of study treatment, patients are followed up at 1, 2, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory B-acute lymphoblastic leukemia (ALL), chronic lymphocytic leukemia (CLL), or non-Hodgkin's lymphoma (NHL) treated with at least two lines of therapy, and have persistent or progressed disease including positive minimal residual disease (MRD)
* Patients may have received last cytotoxic chemotherapy at least 3 weeks prior to lymphodepleting chemotherapy
* Patient may continue targeted therapy until 2 weeks before initiation of lymphodepleting chemotherapy with the exception of ibrutinib
* Disease must be CD19 and/or CD22 positive by flow cytometry or immunohistochemistry
* Karnofsky/Lansky performance scale > 70
* Total bilirubin less than < 1.5 mg/dL except patients with Gilbert syndrome whose total bilirubin must be < 3.0mg/dL
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) =< 2.5 X upper limit of normal (ULN)
* Alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 5.0 ULN
* Serum creatinine (as estimated by Cockcroft Gault) >= 60 cc/min
* Cardiac ejection fraction >= 50% without evidence of pericardiac effusion as determined by echocardiogram (ECHO) or multigated acquisition scan (MUGA), no clinical significant electrocardiogram (ECG) findings
* No clinical significant pleural effusion and baseline oxygen saturation >= 92%
* Absolute lymphocyte count >= 100/ul
* Be able to sign informed consent
* All participants who are able to have children must practice effective birth control while on study. Acceptable forms of birth control for female patients include: birth control pills, patches, or injections, intrauterine device (IUD), diaphragm with spermicide, or condom with spermicide. Acceptable forms of birth control for male patients include condom with spermicide. If female participant becomes pregnant during the study, she will be taken off this study. If male participant fathers a child while on study, he must immediately notify his doctor
* For patients with history of allogenic stem cell transplantation

  * Should not have active acute graft-versus-host disease (GVHD) grade >= 2
  * Should not be on immunosuppressants such as tacrolimus, sirolimus, cyclosporine, mycophenolates for a minimum of a month from CD19-CD22 CAR T cell infusion
  * Should not be on more than physiologic dose of systemic steroid for adrenal insufficiency (prednisone equivalent 5mg/day)
  * Transplantation should be more than 2 months from CD19-CD22 CAR T cell infusion
  * Other cell therapy including CAR T cells, donor lymphocyte infusion, virus specific T cells, natural killer (NK) cells, etc should have 6 weeks of wash-out period from the CD19-CD22 CAR T cell infusion
* For patients with history of central nervous system (CNS) disease, CNS disease must be treated prior to enrollment
* For patients with prior treatment history of cell therapy such as other CAR T cells or CAR NK cells or NK cells, cell therapy should have a 6 weeks of wash-out period from CD19-CD22 CAR T cell infusion
* Be able to consent long-term follow-up protocol PA17-0483

Exclusion Criteria:

* Positive beta-human chorionic gonadotropin (hCG) in female of child bearing potential defined as not postmenopausal for 24 months or no previous surgical sterilization or lactating females
* Known positive serology for human immunodeficiency virus (HIV)
* Presence of active grade 3 or greater toxicity from the previous treatment
* Presence of active fungal, bacterial, viral, or other infection requiring IV antibiotics for management
* Presence of active neurologic disorders
* Concomitant use of other investigational agents
* Current use of corticosteroid more than physiological dose for adrenal insufficiency (prednisone equivalent at a dose higher than 10 mg/day)
* Presence of active CNS disease

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Optimal chimeric antigen receptor (CAR) T cell dose level | Up to 30 days
  Dose-finding will be done using the sequentially adaptive phase I-II EffTox method.
Incidence of adverse events (adverse events) | Up to 30 days
  Toxicity is defined as a grade 3, 4, or 5 cytokine release syndrome, neurotoxicity, or National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 with onset within 30 days of cell infusion. Adverse events that are considered disease-related (not suspected of relationship to CD19-CD22 -CAR T cells) will not be considered dose-limiting toxicities. Only those AEs that occur during the first 30 days after infusion, which are suspected to be related to conditioning lymphodepletion chemotherapy regimen and/or CD19 -CD22-CAR T cells (any component of the treatment regimen), and meet the following criteria, will be used in the definition of toxicity. Hematologic toxicities will not be considered in the definition of toxicity, as pancytopenia is a common toxicity with this regimen.
Efficacy in complete response (CR) or partial response | Day 30 post cell infusion
  Efficacy is defined as the patient being alive and in complete response (CR) or partial response (PR) at day 30 post cell infusion.

SECONDARY OUTCOMES:
Progression-free survival | Up to 1 year post T-cell infusion
  Unadjusted distributions of the time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and T-cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Overall survival | Up to 1 year post T-cell infusion
  Unadjusted distributions of the time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and T-cell dose level will be evaluated by Bayesian piecewise exponential survival regression.

OTHER OUTCOMES:
Immune reconstitution | Up to 1 year post T-cell infusion
  These longitudinal values will be evaluated graphically and cross-tabulated with dose.
Persistence of CAR T-cells | Up to 1 year post T-cell infusion
  These longitudinal values will be evaluated graphically and cross-tabulated with dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jin S Im, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org